CLINICAL TRIAL: NCT06325371
Title: Italian Multicentric Study on the Treatment of Visceral Aneurysms With the Flow Diversion Stent Derivo Peripher and Derivo 2
Acronym: DEDICATE
Status: Recruiting | Type: Observational
Sponsor: University of Turin, Italy (Other)
Responsible Party: Sponsor
Other Study IDs: 0028201
Record Dates: First submitted 2024-03-05; First posted 2024-03-22 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Aneurysm Abdominal; Arterial Aneurysm
Keywords: flow diverter; visceral aneurysm; stenting
MeSH Terms: conditions — Aortic Aneurysm, Abdominal | interventions — Stents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Visceral aneurysm stenting — Flow diverter stenting
  Other Names: stent

SUMMARY:
This is a multicentric voluntary observational study with a retrospective evaluation of prospectively collected data concerning the treatment of visceral aneurysms with flow diversion stent Derivo Peripher and Derivo 2 (DED, Acandis GmbH) Follow-up will include clinical and radiological (CT) evaluation at least 12 months after the intervention.

The enrollment period will be of 65 months (01/jan/2020-30/jun/2025). Sample size will be of 100 patients.

ELIGIBILITY:
Inclusion criteria:

* >18 years old
* Visceral artery aneurysms, evaluated with computed tomography angiography-CTA- withindication for treatment according to 2020 SVS and 2024 SICVE/SIRM and 2024 CIRSE guidelines. Specifically:

  * Renal artery: >2 cm if fusiform morphology or all dimensions if sacculary or bifurcation morphology, if in fertile women or in hypertensive patients with renal stenosis
  * Splenic artery: if >2 cm, or all dimensions in fertile women.
  * Celiac tripod: if >2 cm.
  * Hepatic artery: if >2 cm or growth greater than 0.5 cm/year.
  * Superior mesenteric artery, gastric or gastroepiploic artery, pancreaticoduodenal or gastroduodenal arteries, colic arteries, jejunal arteries, and ileal arteries: any size
* anatomical characteristics compatible with the stent DED Instruction for Use (IFU). Specifically:

  * the stent diameter should match the largest diameter of either the proximal or distal vessel of the aneurysm with an oversizing of 1-2 mm according to IFU.
  * the stent length must allow for adequate proximal and distal landing, covering the neck of the aneurysm to 2.5 times the vessel's internal diameter and no less than 15 mm.
* proper adherence to the anticoagulant and antiplatelet pharmacological protocol for the peri-procedural and post-procedural periods. Specifically:

  * all patients should begin dual antiplatelet therapy (DAPT) before surgery (for at least 3 days before the procedure or with a loading dose pre-procedurally).
  * all patients receive systemic anticoagulation during the procedure (Heparin 70 IU/kg to achieve an Activated Clot Time (ACT) > 250 s).
  * after the procedure, the patient should continue DAPT (e.g., ASA 100 mg daily and Clopidogrel 75 mg daily) for at least 1 month, then continue with single antiplatelet therapy (e.g., ASA 100 mg) indefinitely.

Exclusion Criteria:

* patients who are hemodynamically unstable or show CT signs of rupture or contained rupture of visceral aneurysm
* pregnant or breastfeeding women
* life expectancy less than 2 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men and women >18 years old with the presence of a visceral aneurysm.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-11-20 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Efficacy of the stenting in terms of patency and side branches | 12 months
  stent patency and side branches (the absence of stenosis greater than 50% of the stent's internal lumen and the side branches' lumen)
Efficacy of the stenting in terms of aneurysm thrombosis rate | 12 months
  aneurysm (partial or complete, >50% or 100%) thrombosis
Efficacy of the stenting in terms of aneurysm volume assessment | 12 months
  aneurysm volume assessment (percentage of volume reduction respect to the initial volume)
Safety in terms of morbidity | 12 months
  morbidity (any adverse events occured during follow up for any causes and by causes associated with treatment)
Safety in terms of mortality | 12 months
  mortality (any cause of death related to pathology or not)
Safety in terms of technical issues | 12 months
  technical issues (any adverse event during stent placement)

CONTACTS AND LOCATIONS:
Overall Officials: Marco Calandri, M.D., Principal Investigator — University of Torino
Locations (1):
- AOU Città della Salute e della Scienza di Torino, Torino, TO, Italy

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared to other researchers

REFERENCES:
- [Derived] Discalzi A, Nardelli F, Ficara B, Comelli S, de Donato G, Fanelli F, Quaretti P, Sallemi C, Semeraro V, Sirovich R, Calandri M; DEDICATE Investigators. Study Protocol DEDICATE: Italian Multicenter Study on the Treatment of Visceral Aneurysms with the Derivo Peripher and Derivo 2 Flow Diverter Stent. Cardiovasc Intervent Radiol. 2025 May;48(5):694-701. doi: 10.1007/s00270-025-04016-8. Epub 2025 Mar 13. PMID 40082273